CLINICAL TRIAL: NCT01087775
Title: Enhancing Cognitive Function and Reintegration in Iraq and Afghanistan Veterans With PTSD Using Computer-Based Cognitive Training
Brief Title: GAME Veterans With PTSD Using Computer-Based Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Seal (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Karen Seal, Principle Investigator, San Francisco Veterans Affairs Medical Center
Organization: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH1020078; NCT01552278 (obsolete NCT alias)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive Training (Experimental): Plasticity Based Adaptive Cognitive Remediation (PACR)
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Cognitive Training — Plasticity Based Adaptive Cognitive Remediation (PACR)
  Other Names: Plasticity Based Adaptive Cognitive Remediation (PACR)

SUMMARY:
The investigators hypothesis are as follows:

H1a: OEF/OIF veterans with PTSD who perform cognitive training (CT) will demonstrate greater objective improvements on standard (untrained) neurocognitive measures, with the largest gains in verbal memory, learning and sustained attention.

H1b: Objective cognitive improvements in CT participants will be sustained at three months post-intervention, suggesting persistence of neuroplasticity-based cognitive training benefits.

H2a: OEF/OIF veterans with PTSD who perform CT will report greater improvements in cognitive function.

H2b: OEF/OIF veterans with PTSD who perform CT will demonstrate improved social and occupational functioning and quality of life.

H2c: OEF/OIF veterans with PTSD who perform CT will demonstrate greater improvements in community reintegration.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD)-related cognitive dysfunction is well-described and has been associated with specific impairments in verbal memory, learning, attention and emotional regulation, deficits which have been correlated with abnormalities in specific brain regions. Both PTSD and cognitive dysfunction have been associated with impairments in social and occupational functioning and may contribute to operational or battlefield errors, soldiers' safety and threaten the success of military operations. In addition, following military service separation, PTSD-related cognitive impairment adversely impacts quality of life, readjustment, and community reintegration. A computerized neuroplasticity-based auditory cognitive training program (Plasticity-Based Adaptive Cognitive Remediation, Posit Science, San Francisco, CA) has been shown in several randomized controlled trials to improve verbal memory, attention, cognitive control, quality of life and daily function in community-dwelling elders and individuals with schizophrenia. To our knowledge however, there have been no studies of cognitive remediation training in individuals with PTSD. Therefore, the overall aim of this proposal was to investigate the efficacy of neuroplasticity-based auditory cognitive training in Veterans with PTSD and cognitive dysfunction. The primary specific aim of this pilot study was to examine change in objective cognitive function in Veterans with PTSD and cognitive dysfunction who participated in an open-label trial of an auditory cognitive training program. Our secondary aim was to examine change in self-reported cognitive function, social and occupational functioning, quality of life and community reintegration in Veterans with PTSD who participate in auditory CT. Finally, we evaluated the feasibility and usability of home-based computerized auditory cognitive training in Veterans with PTSD and cognitive dysfunction. We enrolled subjects in a program of 3 months of auditory cognitive training (CT) followed by 3 months of no contact. We assessed participants' change scores on neuropsychological outcome measures from pre- to post-treatment using reliable change indicators. We utilized qualitative thematic analysis to identify themes from participants about the feasibility, acceptability, and usability of the treatment. Information derived from this pilot study may be used to inform future cognitive training interventions for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* An experienced clinical interviewer with Master's-level training will conduct first- and second-level screening to determine study eligibility for enrollment in the randomized controlled trial.
* The First-Level Eligibility Screen will be conducted by phone and will apply the following inclusion criteria in an effort to recruit a homogeneous sample:

  1. Confirmed OEF and/or OIF military service
  2. Male veterans, ages 18 to 40 years with 12 to 16 years of education
  3. History of a prior positive PTSD screen or diagnosis either by SFVAMC study referral or self-report'
  4. Able and willing to travel to SFVAMC
  5. Able and willing to perform daily home-based computer exercises for three months.
* The Second Level Eligibility Determination will occur in-person at the SFVAMC of potential participants who have met first-level screening eligibility criteria. Second-level eligibility screening will require signed informed consent (see below) before the second-level screening is conducted. During the second-level eligibility screen, consenting participants will be administered:

  1. The Clinician-Administered PTSD screen (CAPS) and the Mini International Neuropsychiatric Interview (MINI) 29 to assess for Diagnostic and Statistical Manual (DSM)-IV Axis I psychiatric disorders
  2. The VA TBI second-level screen [TBI event history and Neurobehavioral Symptom Inventory (NSI) for cognitive symptoms].30
* To be eligible for enrollment in the randomized controlled, veterans at second-level screening must:

  1. Meet threshold criteria for current full or sub-syndromal PTSD by DSM-IV criteria 31
  2. Report ≥ 1 moderate or severe cognitive symptom(s) on the NSI that interfere(s) with daily function including moderate to severe poor concentration, forgetfulness, difficulty making decisions and slowed thinking.
* Because PTSD is a highly comorbid condition, eligible participants may have other comorbid stable neuropsychiatric disorders, including depression or a history of a mild traumatic brain injury.

Exclusion Criteria:

* The following exclusion criteria will apply to first-level screening:

  1. Poor English comprehension and fluency
  2. Unstable medical condition, injury or disability, including moderate to severe TBI (by self-report) and hearing impairment
  3. Current (or past 60 day) evidence-based PTSD or cognitive remediation therapy; in contrast, stable supportive therapy for PTSD and/or other mental disorders, such as group therapy or on stable psychoactive medication (> 30 days) will be acceptable.
* The following exclusion criteria will apply to second-level screening:

  1. Drug and alcohol dependence and other unstable serious mental illness (e.g. psychosis) (assessed using the MINI)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen H Seal, MD, Principal Investigator — San Francisco VA Medical Center
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment flyers were posted on poster boards and electronic billboards around the SFVAMC; collaborated with other investigators to refer potential participants; utilized social media and created a website. We targeted community-based VA facilities, other Veteran community based organizations and local colleges and universities.
Period: Overall Study
Arm/Group | Cognitive Training
Started | 25
Completed | 23 (2 subjects were found to be ineligible for the study)
Not Completed | 2
Not completed — failed inclusion criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cognitive Training
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.73 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change Scores of Standard (Untrained) Neurocognitive Measures (Verbal Memory, Learning and Sustained Attention)
Description: We presented change scores (6-month scores minus baseline scores) outcomes of 10 measures of neurocognitive measures (together with ranges): the Wechsler Memory Scale (WMS-IV) Paired Associates immediate and delayed memory (range: 1-19), Rey Auditory Verbal Learning Test (RAVLT) total score (range: 0-100) and delayed score (range: 0-20), Wechsler Adult Intelligence Scale (WAIS-IV) Digit Span (range: 0-48), Wechsler Adult Intelligence Scale (WAIS-IV) Letter Number Sequencing (range: 1-19), Auditory Consonant Trigrams (ACT) raw score (range: 0-60), Delis-Kaplan Executive Function System (D-KEFS) Stroop Inhibition (range: 1-19), and the Brief Visual Memory Test revised (BVMT-R) total T score and Delayed T score (range: 20-80). Higher scores mean better cognitive functioning outcomes.
Time Frame: 6-month follow-up
Population: Challenges in recruitment/retention led us to redesign the study as an open trial and the limitation is that there is a small number of subjects who completed the study.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Treatment: Treatment Arm
Arm/Group | Treatment
Number analyzed (Participants) | 7
score on a scale
  WMS-IV Paired Associates Scaled score | 2.29 [-1 to 6]
  WMS-IV Paired Associates Delayed Scaled score | 2.29 [0 to 6]
  RAVLT Total raw score | 0.71 [-4 to 7]
  RAVLT Delayed raw score | 0.14 [-3 to 3]
  WMS-IV Digit Span Scaled score | 2.43 [0 to 4]
  WMS-IV Letter Number Sequencing scaled score | 0.286 [-1 to 2]
  ACT Raw score | 10.57 [0 to 30]
  D-KEFS Stroop Inhibition Standard score | 2.71 [0 to 9]
  BVMT Total T score | 0.71 [-19 to 29]
  BVMT Delayed T score | 7 [-15 to 34]

2. Secondary Outcome: Social and Occupational Functioning and Quality of Life Scores at 6 Months
Description: To measure social and occupational functioning, we used the World Health Organisation Quality of Life Assessment (WHOQOL-BREF) validated to detect intervention-related change in quality of life.
  Range of post-treatment domain scores:
  WHOQOL physical domain: 7-35; WHOQOL psychological domain: 6-30; WHOQOL social relationships domain: 2-10; WHOQOL environment domain: 8-40.
  Higher scores indicate better quality of life outcomes.
Time Frame: 6 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 7
score on a scale
  WHOQOL physical domain score | 12.65 (2.75)
  WHOQOL psychological domain score | 10.10 (2.29)
  WHOQOL social relationships domain score | 12.76 (3.16)
  WHOQOL environment domain score | 14.00 (2.75)

ADVERSE EVENTS:
Arm/Group | Cognitive Training
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No